CLINICAL TRIAL: NCT02597244
Title: Effectiveness of Percutaneous Foraminotomy in Patients With Lumbar Foraminal Stenosis: A Prospective, Pilot Study
Brief Title: Effectiveness of Percutaneous Foraminotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: BioSpine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sangchul Lee, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0620141940
Record Dates: First submitted 2015-10-06; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Stenosis
Keywords: Lumbar foraminal stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): Percutaneous Extraforaminotomy using BS extraforamonotomy kit(BioSpine Co.,Ltd, Seoul, South Korea)
  Interventions: Device: Percutaneous Extraforaminotomy

INTERVENTIONS:
Device: Percutaneous Extraforaminotomy — percutaneous dissecting of the lumbar extraforaminal and foraminal region with BS extraforamonotomy kit(BioSpine Co.,Ltd, Seoul, South Korea) under fluoroscopy

SUMMARY:
Percutaneous Extraforaminotomy using BS extraforamonotomy kit(BioSpine Co.,Ltd, Seoul, South Korea), was performed in patients who did not show improvement lasting more than 1 month after diagnostic conventional fluoroscopically guided transforaminal epidural block with local anesthetic and steroid.

Numeric rating scale(NRS) pain score, Oswestry disability index (ODI), Roland-Morris Disability Questionnaire (RDQ), claudication distance(CD) was checked before and after the procedure.

DETAILED DESCRIPTION:
Percutaneous Extraforaminotomy with Transforaminal Adhesiolysis may be an effective minimal invasive technique in patients not responsive to conventional epidural steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* radicular pain with positive provocation factors > 3 months
* Radicular pain at L4 or L5
* Presence of dominant side when bilateral symptom present
* Positive provocation factors: leg symptoms elicited or aggravated by walking but relieved by sitting down
* Not appropriate relief of pain routinely conservative treatment (physiotherapy, exercise, analgesic medication, epidural steroid injection) > 3 months
* Magnetic resonance imaging(MRI) : Foraminal stenosis of Grade 1-3 (foraminal herniated intervertebral disc(HIVD) with mild to severe degree of foraminal stenosis according to AJR:194, April 2010 by Lee, et. Al)
* Subjects who signed for the consent form

Exclusion Criteria:

1. Acute back or leg pain
2. Sings of progressive neurologic deficits, including muscle atrophy and abnormal tendon reflexes
3. Patients with a history of prior spine surgery
4. Allergic response to steroid or contrast dye
5. Bleeding diathesis or over coagulopathy
6. Patients with bilateral radiculopathy or spinal stenosis at more than 3 levels

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
NRS score | 4 weeks after intervention
  A comparison of the mean difference in the change of NRS scores of their leg pain from entry to the scores at 4-week

SECONDARY OUTCOMES:
NRS score | 8, 12 weeks after intervention
  A comparison of the mean difference in the change of NRS scores of their leg pain from entry to the scores at 8, 12-weeks after intervention
Oswestry disability index(ODI) | 4, 8 and 12 weeks after intervention
  A change of ODI over periods of time after intervention (12 weeks)
5-point satisfaction scale | 4, 8 and 12 weeks
  Patient satisfaction with treatment at 4, 8, & 12 weeks
Any adverse events | Throughout the study period (up to 12 weeks)
Roland-Morris Disability Questionnaire(RDQ) | 4, 8 and 12 weeks after intervention
  A change of RDQ change over periods of time after intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sangchul Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Result] Cooper G, Lutz GE, Boachie-Adjei O, Lin J. Effectiveness of transforaminal epidural steroid injections in patients with degenerative lumbar scoliotic stenosis and radiculopathy. Pain Physician. 2004 Jul;7(3):311-7. PMID 16858467